CLINICAL TRIAL: NCT03349554
Title: An Exploratory Study of the Feasibility of the Installation by a Paramedical Staff of a Standardized Meditation Technique "Body-scan", in the Management of Anxiety in Hospitalized Parkinsonian Patients
Brief Title: A Standardized Meditation Technique "Body-scan", in the Management of Anxiety in Hospitalized Parkinsonian Patients
Acronym: PARAM2A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2016/50
Record Dates: First submitted 2017-10-26; First posted 2017-11-21 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2018-03

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; anxiety; meditation; in-patients
MeSH Terms: conditions — Parkinson Disease; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- standardized meditation technique "body-scan" (Experimental)
  Interventions: Other: body-scan meditation; Diagnostic Test: Psychological evaluation

INTERVENTIONS:
Other: body-scan meditation — 15 minutes audio-guided body-scan meditation
Diagnostic Test: Psychological evaluation — NPI (Neuropsychiatric symptoms Inventory) - PAS (Parkinson's disease Anxiety Screening Questionnaire) - VAS measuring pain, anxiety and discomfort Before and after "body-scan" meditation

SUMMARY:
The aim of the study is to constitute a proof of concept study for a larger study investigating the effect of mindfulness on anxiety and agitation in Parkinson's disease (PD) based on the results of a preliminary feasibility.

DETAILED DESCRIPTION:
Neuropsychiatric and behavioral non motor symptoms are common in PD often requiring hospitalization and/or specific drug management. Mindfulness-based stress reduction (MBSR) programs have proved to be efficacious in PD both for the management of motor and non-motor symptoms. This is however the case only in out-patients and by using standardized 8 weeks programs. The team has experienced in the hospitalization unit that methods derived from the MBSR program such as the "body scan", administered by the paramedical personnel, is of great help for the non-pharmacological management of anxiety and agitation in PD, avoiding physical contention in many cases. Based on this experience the study aims at evaluating the feasibility and preliminary efficacy of a simple and standardized administration of the "body scan" meditation in the management of anxiety and agitation in PD admitted in the unit since less than 48h.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease
* Age over 18
* Admitted in the unit since less than 3 days
* Presenting at least 3 symptoms with a severity rated > 2 at the Hamilton anxiety scale (HAM-A)
* Patients with social security insurance
* Informed consent signed

Exclusion Criteria:

* Dementia, delusions or hallucination not permitting an informed consent or necessitating immediate and urgent sedation
* Patient under law protection
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-03-05 (Actual)

PRIMARY OUTCOMES:
Percentage of patients that received a first experience of standardized "body scan" meditation within 48H after admission | 48 hours after admission

SECONDARY OUTCOMES:
Rate of patient's eligibility and causes of non-eligibility | At inclusion (day 0)
Rate of study drop-out | through study completion, an average of 1 year
Causes of study drop-outs | through study completion, an average of 1 year
  by oral questionnaire
Mean delay between admission and first meditation | After "body scan" meditation, an average of 48 hours after admission
Cause of failure of meditation administration within 48h | 48 hours after admission (day 0)
  Failure factors: related to staffing (insufficient, untrained...), related to the organization of the service (double room / individual), related to the patient (visits, temporary refusal), related to the equipment (unavailable, non-functional)
Percentage of improvement pain, anxiety and discomfort | before and after "body scan" meditation, an average of 48 hours after admission
  by visual analog scales (VAS)
Percentage of improvement at the Parkinson's disease | before and after "body scan" meditation, an average of 48 hours after admission
  by Anxiety Screening Questionnaire (PAS)
Percentage of improvement at the Parkinson's disease | before and after "body scan" meditation, an average of 48 hours after admission
  by the Neuropsychiatric symptoms Inventory (NPI) total scores

CONTACTS AND LOCATIONS:
Overall Officials: François TISON, Prof, Study Director — University Hospital Bordeaux, France; Caroline GAUTIER, Principal Investigator — University Hospital Bordeaux, France
Locations (1):
- Service de neurologie motricité,Hôpital Pellegrin, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No